CLINICAL TRIAL: NCT03697889
Title: An Open-label, Randomized, Single-dose, Two-treatment, Crossover Bioequivalence Study Comparing a Novel Naproxen Sodium 275 mg Film-coated Tablet (BILIM ILAC SANAYII VE TICARET A.S., TURKEY) and Nalgesin® 275 mg Naproxen Sodium Film-coated Tablet (JSC "KRKA, D.D., NOVO MESTO", SLOVENIA), in Healthy Adult Volunteers
Brief Title: A Study to Assess Bioquivalence Between a Novel Naproxen Sodium 275 mg Film-coated Tablet and Nalgesin Naproxen Sodium 275 mg Film-coated Tablet in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CO-171115092223-PACT
Record Dates: First submitted 2018-10-04; First posted 2018-10-05 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Healthy
Keywords: Bioequivalence
MeSH Terms: interventions — Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence AB (Experimental): Participants will receive Treatment A (test product Naproxen sodium tablet, 1 x 275 mg) at dosing period 1 followed by Treatment B (reference product Nalgesin, 1 x 275 mg) dosing period 2. There is a wash-out period of 7 days between the two dosing periods.
  Interventions: Drug: Naproxen sodium (test product); Drug: Naproxen sodium (reference product)
- Treatment Sequence BA (Experimental): Participants will receive Treatment B (reference product Nalgesin, 1 x 275 mg) at dosing period 1 followed by Treatment A (test product Naproxen sodium tablet, 1 x 275 mg) at dosing period 2. There is a wash-out period of 7 days between the two dosing periods.
  Interventions: Drug: Naproxen sodium (test product); Drug: Naproxen sodium (reference product)

INTERVENTIONS:
Drug: Naproxen sodium (test product) — Participants will be administered single doses of 275 mg Naproxen sodium (test product) tablet orally.
Drug: Naproxen sodium (reference product) — Participants will be administered single doses of 275 mg Naproxen sodium (reference product - Nalgesin) tablet orally.
  Other Names: Nalgesin

SUMMARY:
This is a research study designed to evaluate the rate and extent of absorption of Naproxen from a novel Naproxen sodium tablet and Nalgesin naproxen sodium 275 mg.

DETAILED DESCRIPTION:
The study has an open-label, randomized, two-way crossover design. 28 healthy participants will be included. Single-doses of 1 tablet of Naproxen sodium 275 mg and Nalgesin 275 mg will be given on separate treatment visits to healthy adult participants under fasting conditions. A crossover design is chosen in order to allow within-subject comparisons of treatments. To minimize the risk of carry-over effect, the washout period between the study drug administrations is set to 7 days. The study is open-label because the primary data collected are concentration measurements that cannot be expected to be affected by a participant's knowledge of the product administered.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subject between the ages of 18 and 45 years, inclusive. Healthy is defined as the absence of any disease or abnormalities (including positive test for human immunodeficiency virus (HIV) 1 or 2 antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (anti-HCV) or syphilis (RW)) as judged by the investigator on the basis of a detailed medical history, physical examination, blood pressure, pulse rate measurements, 12-lead electrocardiogram, as well as clinical laboratory tests. The responsible investigator may request additional investigations or analyses if necessary
* Non- or ex-tobacco user, being defined as someone who completely stopped smoking or using any form of tobacco or nicotine-containing product for at least 12 months before 1st dose of the study drug in this study.
* Females: Postmenopausal state (absence of menstrual discharge for at least two years and a follicle stimulating hormone (FSH) serum level exceeding 30 IU/L) or premenopausal/perimenopausal state with an effective means of contraception (oral, injected, implanted, or transdermal hormonal contraceptives, vaginal contraceptive ring, intrauterine device, or status after operative sterilization) during the study and 30 days thereafter, single male partner who has had a vasectomy, or abstinence from heterosexual intercourse, during the study and 30 days thereafter.
* Males: No pregnant spouse or partner at screening and willingness to protect potential spouse or partner from becoming pregnant during the study and 30 days thereafter.
* Body Mass Index (BMI) ≥ 18.5 and ≤ 30.0 kg/m2 with a total body weight >50 kg.
* A personally signed and dated informed consent document, indicating that the subject has been informed of all pertinent aspects of the study.
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures specified in the protocol.

Exclusion Criteria:

* Use of medications other than contraceptives specified in Inclusion criterion 3 or occasional use of other medications approved by the Investigator.
* Use of any vitamins, dietary and herbal supplements within 7 days before each dose of study drugs.
* Use of any nonprescription or prescription medications, including naproxen medications, other than contraceptives, within 5 times the drug's half-life before each dose of study drug.
* Depot injection or an implant of any drug within 3 months prior to dosing.
* History of any allergy or hypersensitivity (e.g. skin reaction, asthma, angioedema) to naproxen, ibuprofen, ASA, other NSAIDs or any related products (including excipients of the formulations).
* Females: Confirmed pregnancy or a positive pregnancy test at the screening visit, or planning to become pregnant during the duration of the study, and/or breast-feeding
* Has a history of peptic ulcers, gastrointestinal bleeding of any etiology, bleeding disorders, gastrointestinal disease (including chronic heartburn or gastroesophageal reflux disease), inflammatory bowel disease (ulcerative colitis, Crohn's disease), or gastrointestinal surgery other than appendectomy.
* Has asthma, hypertension, fluid retention, or heart disease either by history or by the medically qualified principal investigator's medical judgment; has hemophilia and other disorders of blood clotting and hemostasis disorders, has cerebrovascular hemorrhage or other hemorrhages;
* Has renal or hepatic impairment; according to the medically qualified investigator discretion;
* Acute infectious disease within 4 weeks prior to screening.
* Treatment with an investigational drug within 3 months preceding the first dose of study treatment.
* Preplanned surgical procedures during the study period, if this may interfere with the conduct of the study.
* History of alcoholism defined as alcohol consumption in the 6 months before screening that exceeds weekly limits of 10 alcohol units (2 L of wine or 5 L of beer or 0.5 L of spirits) or substance abuse, as judged by the Investigator, within the past 6 months preceding this study.
* Consumed alcohol beverage(s) within 48 hours prior to the first scheduled dose of the study drug, positive respiratory alcohol test at screening, or inability to abstain from alcohol consumption during the entire study period.
* Positive urine screen for drug abuse.
* Use of xanthine containing products (e.g., coffee, tea, chocolate or cola drink) within 48 hours before each dose of study drug.
* Ingestion of food or beverages containing grapefruit, Chinese grapefruit (pomelo) or Seville oranges (including marmalade) within 10 days before the first dose of study drug and throughout the study.
* Donation or loss of blood within 3 months prior to the first dose of study drug if the estimated lost blood volume equaled or exceeded 450 mL.
* Abnormal results of laboratory and instrumental methods of examinations, including electrocardiogram (ECG) at screening;
* Heart rate <60 or >90 per minute at rest, or systolic blood pressure <100 or >130 mm Hg, or diastolic blood pressure <70 or >90 mm Hg measured at screening visit.
* Has any acute or chronic, medical or psychiatric condition(s) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the medically qualified investigator, would make the subject inappropriate for entry into this study;
* Relationship to persons involved directly in the conduct of the study (i.e., principal investigator, subinvestigators,study coordinators, other study personnel, employees or contractors of the sponsor or Johnson & Johnson subsidiaries, and the family of each).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
The maximum observed plasma concentrations (Cmax) of Naproxen Sodium | 15, 30, 45 minutes, and at 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours after drug administration
  The maximum observed plasma concentration (Cmax)
The area under the plasma concentration-vs.-time curves from start of Naproxen sodium administration until the time of the last measurable concentration (AUCt) | 15, 30, 45 minutes, and at 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours after drug administration
  AUCt is defines as area under the plasma concentration versus time curves from start of drug administration until the last measureable concentration.

SECONDARY OUTCOMES:
The area under the plasma concentration-vs.-time curve from the start of Naproxen sodium administration extrapolated to infinity (AUC∞) | 15, 30, 45 minutes, and at 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours after drug administration
  AUC∞ is defined as area under the plasma concentration versus time curves from start of drug administration until the nicotine plasma concentration is negligible (infinity).
The extrapolated part of AUC∞, AUCExtrap | 15, 30, 45 minutes, and at 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours after drug administration
The time at which maximum Naproxen sodium concentraton (Cmax) is observed (Tmax) | 15, 30, 45 minutes, and at 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours after drug administration
  Tmax is defined as the time point at which the maximum nicotine concentration (Cmax) occurs
The terminal elimination rate constant (lambda-z) for Naproxen sodium | 15, 30, 45 minutes, and at 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours after drug administration
  The rate at which the drug is removed from the body system.
The terminal elimination half-life (t1/2) of Naproxen sodium | 15, 30, 45 minutes, and at 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours after drug administration
  The time taken for the Naproxen sodium plasma concentration to fall to half its original value.
Number of participants with Adverse Events | Approximately 26 days
  An AE is any untoward from a medical standpoint event occurred in patient or subject of clinical study after the use of a medicinal product which may or may not have a causal relationship with its use.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin A. Zacharov, MD, Principal Investigator — LLC "Scientific and Research centre Eco-safety"
Locations (1):
- LLC "Scientific and Research centre Eco-safety", Saint Petersburg, Russia

REFERENCES:
- See also: Synopsis to support result registration for a clinical study performed within the Russian federation. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CO-171115092223-PACT&attachmentIdentifier=f8a0d9d8-c13a-4ad7-9ebb-b24720e90711&fileName=Redacted_bluefish_synopsis.pdf&versionIdentifier=